CLINICAL TRIAL: NCT05109247
Title: Prediction of Spontaneous Onset of Labor at Term
Acronym: PREDICT
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: Hologic, Inc. (Industry); QIAGEN Gaithersburg, Inc (Industry); Pregnolia AC (Unknown)
Responsible Party: Principal Investigator, Federico Migliorelli, Obstetrician, Principal Investigator, University Hospital, Geneva
Other Study IDs: 19-261
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Labor, Induced; Labor, Obstetric; Labor Onset; Predictive Model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study intends to develop a predictive model of spontaneous onset of labor between 39 and 41 weeks of pregnancy in women carrying singletons and without indication of delivery before this date. The main hypothesis is that a combination of clinical, ultrasonographic, biochemical and/or biophysical variables will allow to differentiate women who will spontaneously trigger their labors from those who will require an induction by the term of their pregnancies. A tool of this kind should aid in the individualization of the management of the final weeks of pregnancy and, at the light of recent evidence, provide support to the decision-making processes.

ELIGIBILITY:
Inclusion Criteria:

* Alive fetus
* Singletons
* Cephalic presentation
* Intact membranes
* Gestational age ≥ 38 weeks and 5 days

Exclusion Criteria:

* Fetal malformations
* Symptomatic uterine contractions
* Contraindication for vaginal delivery
* Medical indication of induction of labor or elective cesarean delivery
* Maternal desire to induce labor
* Maternal negative to enrollment
* Language barrier
* Inability to give consent

Specific Exclusion Criteria for Pregnolia System (if any of these criteria is present, the measurement of cervical stiffness using Pregnolia aspiration device will not be performed):

* Müllerian anomalies with two cervices
* Severe vaginal bleeding
* Cervical dilatation
* Known HIV
* Visible, symptomatic cervical or vaginal infections
* If one of the following conditions is present on the cervix at the 12 o'clock position:

  * Nabothian cyst
  * Cervical myomas
  * Cervical condylomas
  * Squamous intraepithelial lesion
  * Conization/LEEP2/LLETZ3
  * Cervical endometriosis
  * Cervical tears
  * Cervical dysplasia
  * Large ectopy, for which it is not possible to find a suitable location near the ectopy where native tissue is present
  * Large scar tissue, for which it is not possible to find a suitable location near the scar where native tissue is present.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women at 38+5 - 39 weeks of gestation who will deliver at the centers in which the study will be carried out.
Sampling Method: Non-Probability Sample
Enrollment: 429 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Spontaneous versus induced onset of labor | 3 weeks
  Number of participants who will spontaneously go into labor between the 39th and the 41st week of pregnancy versus number of participants requiring an induction of labor during the 41st week of pregnancy due to advanced gestational age

SECONDARY OUTCOMES:
Gestational age at spontaneous onset of labor | 2 weeks
  Time from sample collection at 39 weeks of pregnancy to spontaneous onset of labor
Gestational age at spontaneous onset of labor | 1 week
  Time from sample collection at 40 weeks of pregnancy to spontaneous onset of labor

CONTACTS AND LOCATIONS:
Locations (3):
- Switzerland (3):
  - Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud
  - Universitätsspital Basel, Basel
  - Hôpitaux Universitaires de Genève, Geneva

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Migliorelli F, Ferrero L, McCarey C, Marcenaro S, Othenin-Girard V, Chilin A, Martinez de Tejada B. Prediction of spontaneous onset of labor at term (PREDICT study): Research protocol. PLoS One. 2022 Jul 13;17(7):e0271065. doi: 10.1371/journal.pone.0271065. eCollection 2022. PMID 35830435